CLINICAL TRIAL: NCT03638817
Title: Evaluation of Perioperative Eltrombopag for the Management of Elective Surgery and Invasive Acts in Patients With Inherited Thrombocytopenia
Brief Title: Perioperative Eltrombopag in Patients With Inherited Thrombocytopenia
Acronym: ELPOT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: French network for inherited hemorragic diseases (Unknown); National Reference Centre for Platelet Pathologies (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/16/8913; 2017-004489-88 (Other: EudraCT Number)
Record Dates: First submitted 2018-06-29; First posted 2018-08-20 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Thrombocytopenia
Keywords: Inherited thrombocytopenias (IT); Platelet concentrates (PC); Eltrombopag; Surgery; Invasive acts; Perioperative; Rare disease; Thrombopoietin mimetic
MeSH Terms: conditions — Thrombocytopenia; Rare Diseases | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eltrombopag (Experimental)
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag will be prescribed at doses recommended in primary immune thrombocytopenia (50, 25 or 75 mg), starting 4 weeks before the procedure and stopped 2 days before. PC will be administrated prophylactically if the platelet count is < 80 G/L or per/post-operatively in case of bleeding of undetermined cause.
  Antifibrinolytics will be authorized and low molecular weight heparin prescribed if indicated for the prophylaxis of postoperative venous thrombosis according to the standard dose and duration, , irrespective of the platelet count

SUMMARY:
The objective of the study is to estimate the response to eltrombopag based on platelet count increase above a safety level of 80 G/L and lack of requirement for pre-, per- and post-operative administration of platelet concentrates (PC) for performing elective invasive acts at mild or high bleeding risk,in selected patients with inherited thrombocytopenia (IT).

DETAILED DESCRIPTION:
The hypothesis of the trial is that preoperative treatment by a thrombopoietin mimetic (eltrombopag) will be effective and safe and will avoid requirement of PC administration in a majority of IT patients Eltrombopag is a thrombopoietin mimetic available orally, not licenced for the treatment of IT. Preliminary data in short series of IT patients indicate that eltrombopag, at the doses used in primary immune thrombocytopenia, increases the platelet counts after 2-4 weeks of treatment and reduces spontaneous bleeding in a significant proportion of subjects. The tolerance of short-term treatment is good. The experience of eltrombopag for the management of perioperative thrombocytopenia in IT is anecdotic. Avoiding the administration of platelet concentrates in these patients, especially children, would represent a direct benefit by preventing adverse reactions to transfusion of blood products and human leukocyte antigen (HLA) immunisation.

Eltrombopag will be prescribed after the inclusion visit at the standard dose of 50 mg/day with dose adjustment on the platelet count (+/- 25 mg) after 2 weeks, for a maximum of 4 weeks before the invasive procedure. If the predefined safety level of platelet count required for the procedure is reached, the treatment will be discontinued and the patient operated without prophylactic administration of PC. In case of bleeding of undetermined cause per-and post-operatively, rescue PC will be given.

Clinical and biological follow-up will be performed until the end-of-study visit, 4 weeks after the intake of the last tablet of eltrombopag.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients with bleeding history and chronic thrombocytopenia with strong presumption of constitutional origin on the basis of

  * the identified mutation and/or
  * a combination of the following criteria: familial antecedent with Mendelian transmission, duration of thrombocytopenia, suggestive syndromic presentation, and evidence against primary or secondary immune thrombocytopenia, especially absence of immunologic markers and failure of previous conventional or immunosuppressive therapies.
* Averaged platelet counts during the last five years below the safety level required for the procedure.
* Scheduled (>4 weeks) surgery or invasive procedure with anticipated risk of bleeding: e.g. needle biopsy of solid organ (liver, kidney….etc.), interventional endoscopy, major surgeries, or surgery without possibility of mechanical control of haemostasis (e.g. tonsillectomy). Written informed consent of the patient or his (her) parents or tutors (patients < 18 yrs).

Patients included in the French national registry of rare platelet disorders

* Patient with social insurance coverage

Exclusion Criteria:

* questionable constitutional origin;
* definite platelet dysfunction associated to thrombocytopenia (eg: gray platelet syndrome, NBEAL2 and related gene mutations, homozygous Bernard-Soulier Syndrome);
* thrombocytopenia with predisposition to hematologic malignancies (e.g; RUNX1, ETV6 or ANKRD26 gene mutations).
* amegakaryocytic thrombocytopenia resulting from mutations in the thrombopoietin (TPO) TPO-Mpl receptor, supposed, by definition, to be hardly responsive to receptor agonists.
* questionable requirement of prophylactic PC transfusions;
* procedure usually associated with platelet consumption requiring transfusions of PC (e.g.: cardiac surgery), making difficult the evaluation of success or failure;
* procedures at risk of bleeding with immediate vital or functional consequences (e.g.: intra cranial surgery);
* personal history of arterial or venous thromboembolic events or known familial thrombophilia;
* association with another acquired or constitutional hemorrhagic diathesis;
* chronic hepatitis, cirrhosis, with moderate to severe liver failure (Child-Pugh score ≥5);
* previous or concurrent myeloid malignancy, including myelodysplastic syndrome;
* alanine aminotransferase (ALT) or bilirubin levels 2 times the upper limit of normal (ULN);
* altered renal function (creatinin clearance <30 ml/min);
* pregnancy (negative test required before inclusion in fertile women) or lactating women;
* refusal of safe contraception;
* ocular lenses opacity;
* hypersensitivity to eltrombopag or one of excipients;
* previous participation to the present study;
* current treatment with antiplatelet drugs, anticoagulants or direct acting antiviral agents approved for treatment of chronic hepatitis C infection;
* psychiatric, social or behavioral condition judged to be non-compatible with the respect of the protocol, including good observance of treatment and compliance to follow-up;
* adult protected by the law.

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Perioperative management by eltrombopag in inherited thrombocytopenia | up to 4 weeks after completion of treatment
  The response to Eltrombopag is a composite criteria including the level of platelet count 2 days before the procedure and the requirement of PC administration at any time in the study period. The "study period" is running from the start of treatment (inclusion visit) to 4 weeks after completion of treatment. A platelet count remaining below 80 G/L preoperatively, whether or not eltrombopag was taken, is a criterion of failure of treatment.

SECONDARY OUTCOMES:
Adverse events | up to 4 weeks after completion of treatment
  Adverse events and adverse reactions occurring at any time during the study period will be collected. Adverse events may be clinical and biological (especially liver function tests).
Excessive bleeding | up to 4 weeks after completion of treatment
  Excessive or unusual bleeding occurring at any time during the study period are major adverse events. An independent event adjudication committee (EAC) will review all bleeding events.
Vascular thrombosis | up to 4 weeks after completion of treatment
  Symptomatic thrombosis (venous or arterial) occurring at any time during the study period will be diagnosed by appropriate objective methods and reviewed by the EAC.
Doses of eltrombopag on-treatment | 2 and 4 weeks after the beginning of the treatment
  The total doses of eltrombopag given in the preoperative period will be recorded, as the dose and duration of treatment required to obtained the safety level
Platelet kinetics | up to 4 weeks after completion of treatment
  Serial blood sampling during the study period will be performed for measuring the rise of platelet count on-treatment and its decline after completion of treatment.
Platelet size | Inclusion and before the procedure
  Mean platelet volume will be measured by flow cytometry.on blood samples obtained for platelet counts at inclusion, during hospitalisation and end-of study visit
Baseline of Serum Thrombopoietin | Inclusion visit
  Serum thrombopoietin will be measured once, at the inclusion visit.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre SIE, Prof., Principal Investigator — University Hospital, Toulouse
Locations (25):
- France (25):
  - Angers Hospital, Angers
  - Bensancon Hospital, Besançon
  - Bordeaux Hospital, Bordeaux
  - Caen Hospital, Caen
  - Clermont-Ferrand Hospital, Clermont-Ferrand
  - Dijon Hospital, Dijon
  - Lille Hospital, Lille
  - Hospices Civils Lyon, Lyon
  - Marseille Hospital, Marseille
  - Montpellier Hospital, Montpellier
  - Nancy Hospital, Nancy
  - Nantes Hospital, Nantes
  - Cochin Hospital, Paris
  - Hopital Europeen G Pompidou, Paris
  - Kremlin Bicetre Hospital, Paris
  - Necker Hospital, Paris
  - Robert Debré Hospital, Paris
  - Trousseau Hospital, Paris
  - Poitiers Hospital, Poitiers
  - Reims Hospital, Reims
  - Rennes Hospital, Rennes
  - Rouen Hospital, Rouen
  - Strasbourg Hospital, Strasbourg
  - university hospital Toulouse, Toulouse
  - Tours Hospital, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pecci A, Gresele P, Klersy C, Savoia A, Noris P, Fierro T, Bozzi V, Mezzasoma AM, Melazzini F, Balduini CL. Eltrombopag for the treatment of the inherited thrombocytopenia deriving from MYH9 mutations. Blood. 2010 Dec 23;116(26):5832-7. doi: 10.1182/blood-2010-08-304725. Epub 2010 Sep 15. PMID 20844233
- [Background] Pecci A. Pathogenesis and management of inherited thrombocytopenias: rationale for the use of thrombopoietin-receptor agonists. Int J Hematol. 2013 Jul;98(1):34-47. doi: 10.1007/s12185-013-1351-7. Epub 2013 May 1. PMID 23636669
- [Background] Pecci A, Barozzi S, d'Amico S, Balduini CL. Short-term eltrombopag for surgical preparation of a patient with inherited thrombocytopenia deriving from MYH9 mutation. Thromb Haemost. 2012 Jun;107(6):1188-9. doi: 10.1160/TH12-01-0005. Epub 2012 Mar 8. No abstract available. PMID 22398565
- [Background] Gerrits AJ, Leven EA, Frelinger AL 3rd, Brigstocke SL, Berny-Lang MA, Mitchell WB, Revel-Vilk S, Tamary H, Carmichael SL, Barnard MR, Michelson AD, Bussel JB. Effects of eltrombopag on platelet count and platelet activation in Wiskott-Aldrich syndrome/X-linked thrombocytopenia. Blood. 2015 Sep 10;126(11):1367-78. doi: 10.1182/blood-2014-09-602573. Epub 2015 Jul 29. PMID 26224646
- [Background] Favier R, Feriel J, Favier M, Denoyelle F, Martignetti JA. First successful use of eltrombopag before surgery in a child with MYH9-related thrombocytopenia. Pediatrics. 2013 Sep;132(3):e793-5. doi: 10.1542/peds.2012-3807. Epub 2013 Aug 12. PMID 23940247
- [Background] Fiore M, Saut N, Alessi MC, Viallard JF. Successful use of eltrombopag for surgical preparation in a patient with ANKRD26-related thrombocytopenia. Platelets. 2016 Dec;27(8):828-829. doi: 10.1080/09537104.2016.1190446. Epub 2016 Jun 8. No abstract available. PMID 27276516
- [Background] Zhang J, Liang Y, Ai Y, Xie J, Li Y, Zheng W. Thrombopoietin-receptor agonists for children with immune thrombocytopenia: a systematic review. Expert Opin Pharmacother. 2017 Oct;18(15):1543-1551. doi: 10.1080/14656566.2017.1373091. Epub 2017 Sep 4. PMID 28845713